CLINICAL TRIAL: NCT03417921
Title: A Randomized Phase I/II Open Label Study to Assess the Efficacy and Safety of ABTL0812 in Combination With Gemcitabine and Nab-paclitaxel in Patients With Advanced Metastatic Pancreatic Cancer at First Line Therapy
Brief Title: A Study of ABTL0812 in Pancreatic Cancer
Acronym: Pancreatic
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We opened another study.
Sponsor: Ability Pharmaceuticals SL (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-C6-2017
Record Dates: First submitted 2018-01-22; First posted 2018-01-31 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ABTL0812; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): ABTL0812 (starting 1,300 mg tid orally) in combination with gemcitabine and nab-paclitaxel will be administered to patients with pancreatic cancer
  Interventions: Drug: ABTL0812; Drug: Gemcitabine and nab-paclitaxel
- ARM B (Active Comparator): Gemcitabine and nab-paclitaxel will be administered to patients with pancreatic cancer as standard pattern
  Interventions: Drug: Gemcitabine and nab-paclitaxel

INTERVENTIONS:
Drug: ABTL0812 — ABTL0812 in combination with gemcitabine and nab-paclitaxel
  Arms: ARM A
Drug: Gemcitabine and nab-paclitaxel — Gemcitabine and nab-paclitaxel as standard pattern

SUMMARY:
A Randomized Phase I/II Open Label Study to Assess the Efficacy and Safety of ABTL0812 in Combination With Gemcitabine and Nab-paclitaxel in Patients With Advanced Metastatic Pancreatic Cancer at First Line Therapy.

DETAILED DESCRIPTION:
This is an open-label, randomized phase I/II multicenter study to evaluate ABTL0812 in combination with gemcitabine and nab-paclitaxel at first line therapy. Patients will be assigned to the following groups during the study conduct:

* GROUP A: You will receive the standard treatment of chemotherapy and the investigational drug ABTL0812.
* GROUP B: You will receive the standard treatment of chemotherapy.

For GROUP A:

Phase I: A 3+3 de-escalation design followed by an expansion phase will be performed

* ABTL0812 will be administered chronically daily. Potential dose levels are 1300 mg tid, 1000 mg tid, 650 mg tid and 500 mg tid. Intrapatient escalation or de-escalation is not permitted. A run-in period of one week for ABTL0812 is planned before starting the first cycle of chemotherapy.
* Chemotherapy will be administered on 28-day cycles: gemcitabine 1000 mg/m2 + nab-paclitaxel 125 mg/m2 on days 1, 8 and 15.
* If any, or all, the components of the chemotherapeutic regimen must be interrupted for any reason (excluding disease progression), ABTL0812 will be administered as maintenance therapy until disease progression, onset of unacceptable drug toxicities, or patient/physician's request to discontinue.

Phase II:

* ABTL0812 will be administered chronically daily at the Recommended Phase 2 Dose (RP2D). A run-in period of one week for ABTL0812 is planned before starting the first cycle of chemotherapy.
* Chemotherapy will be administered on 28-day cycles: gemcitabine 1000 mg/m2 IV + nab-paclitaxel 125 mg/m2 IV on days 1, 8 and 15
* If any, or all, the components of the chemotherapeutic regimen must be interrupted for any reason (excluding disease progression), ABTL0812 will be administered as maintenance therapy until disease progression, onset of unacceptable drug toxicities, or patient/physician's request to discontinue.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Willing and able to provide informed consent
* Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol
* Patient has histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. The definitive diagnosis of metastatic pancreatic adenocarcinoma will be made by integrating the histopathological data within the context of the clinical and radiographic data. Patients with islet cell neoplasms are excluded. Initial diagnosis of metastatic disease must have occurred ≤6 weeks prior to inclusion in the study.
* Patient has one or more metastatic tumors measurable by CT scan (or MRI, if patient is allergic to CT contrast media).
* Patient has not received previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* Patient has not received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Adequate hematologic function, measured as:

  * absolute neutrophil count ≥ 1.5x109/L
  * platelet count ≥ 100x109/L
  * hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 x ULN
* Albumin ≤ 1.5 x ULN AST (SGOT) ≤ 2.5 times x upper limit of normal (ULN) and ALT (SGPT) < 2.5 times x upper limit of normal (≤5 times the ULN in patients with evidence of liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN (≤5 times the ULN in patients with evidence of liver metastases)
* Serum creatinine ≤1.5 ULN
* Have adequate tumor tissue available (either archival or new tumor biopsy) for biomarker analyses. The most recently collected tumor tissue sample should be provided, if available.
* Life expectancy ≥ 12 weeks in the opinion of the investigator
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 guidelines with at least one "target lesion" to be used to assess response. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented
* Contraception: All female patients will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months' consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically. Female patients of childbearing potential must agree to use two forms of highly effective contraception methods during the study and for a period of 6 months following the last administration of the study drug. Male patients and their female partners, who are of childbearing potential and are not practicing total abstinence, must agree to use two forms of highly effective contraception during the study and for a period of 6 months following the last administration of the study drug.
* Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ grade 1 (as defined by Common Terminology Criteria for Adverse Events version 4.03).

Exclusion Criteria:

Inclusion criteria:

Patients fulfilling the following criteria are eligible for participation in the study:

* Patients ≥18 years of age
* Willing and able to provide informed consent
* Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol
* Patient has histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. The definitive diagnosis of metastatic pancreatic adenocarcinoma will be made by integrating the histopathological data within the context of the clinical and radiographic data. Patients with islet cell neoplasms are excluded. Initial diagnosis of metastatic disease must have occurred ≤6 weeks prior to inclusion in the study.
* Patient has one or more metastatic tumors measurable by CT scan (or MRI, if patient is allergic to CT contrast media).
* Patient has not received previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* Patient has not received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Adequate hematologic function, measured as:

  * absolute neutrophil count ≥ 1.5x109/L
  * platelet count ≥ 100x109/L
  * hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 x ULN
* Albumin ≤ 1.5 x ULN AST (SGOT) ≤ 2.5 times x upper limit of normal (ULN) and ALT (SGPT) < 2.5 times x upper limit of normal (≤5 times the ULN in patients with evidence of liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN (≤5 times the ULN in patients with evidence of liver metastases)
* Serum creatinine ≤1.5 ULN
* Have adequate tumor tissue available (either archival or new tumor biopsy) for biomarker analyses. The most recently collected tumor tissue sample should be provided, if available.
* Life expectancy ≥ 12 weeks in the opinion of the investigator
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 guidelines with at least one "target lesion" to be used to assess response. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented
* Contraception: All female patients will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months' consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically. Female patients of childbearing potential must agree to use two forms of highly effective contraception methods during the study and for a period of 6 months following the last administration of the study drug. Male patients and their female partners, who are of childbearing potential and are not practicing total abstinence, must agree to use two forms of highly effective contraception during the study and for a period of 6 months following the last administration of the study drug.
* Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ grade 1 (as defined by Common Terminology Criteria for Adverse Events version 4.03).

Exclusion criteria:

Patients who meet one of more of the following criteria are not eligible:

* Patients with neuroendocrine tumors or cystic neoplasms are excluded
* Patient has received previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present. Patients having received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting are not eligible for this study
* Patient has only locally advanced disease.
* Patients has symptomatic brain metastases. Patients with asymptomatic brain metastases can be included in the study if they are kept on stable doses of steroids for a period of 1 month prior to study entry provided they don't have peripheric neuropathy grade 2 or superior.
* Patients previously treated with an inhibitor of the PI3K/Akt/mTOR pathway
* Patients has gastrointestinal abnormalities including inability to take oral medications, malabsorption syndromes or other clinically significant gastrointestinal abnormalities that may impair the absorption of the investigational medicinal product.
* Pregnancy or lactation. Serum pregnancy test to be performed within 7 days prior to study treatment start.
* Patients had myocardial infarction within ≤ 12 months prior to study entry, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina pectoris, or unstable cardiac arrhythmia requiring medication.
* Evidence of pre-existing uncontrolled hypertension. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Patients has active Hepatitis B or C or human immunodeficiency virus (HIV) infection with non-controlled disease according to the treating physician.
* Patients with any other medical conditions (such as psychiatric illness, infectious diseases, abnormal physical examination or laboratory findings) that in the opinion of the investigator may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Emergent Adverse Events | 1 year
  Related Adverse Events as Assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Carles Domènech, PhD, Study Director — Ability Pharmaceuticals SL
Locations (1):
- Marc Cortal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erazo T, Lorente M, Lopez-Plana A, Munoz-Guardiola P, Fernandez-Nogueira P, Garcia-Martinez JA, Bragado P, Fuster G, Salazar M, Espadaler J, Hernandez-Losa J, Bayascas JR, Cortal M, Vidal L, Gascon P, Gomez-Ferreria M, Alfon J, Velasco G, Domenech C, Lizcano JM. The New Antitumor Drug ABTL0812 Inhibits the Akt/mTORC1 Axis by Upregulating Tribbles-3 Pseudokinase. Clin Cancer Res. 2016 May 15;22(10):2508-19. doi: 10.1158/1078-0432.CCR-15-1808. Epub 2015 Dec 15. PMID 26671995
- [Background] Munoz-Guardiola P, Casas J, Megias-Roda E, Sole S, Perez-Montoyo H, Yeste-Velasco M, Erazo T, Dieguez-Martinez N, Espinosa-Gil S, Munoz-Pinedo C, Yoldi G, Abad JL, Segura MF, Moran T, Romeo M, Bosch-Barrera J, Oaknin A, Alfon J, Domenech C, Fabrias G, Velasco G, Lizcano JM. The anti-cancer drug ABTL0812 induces ER stress-mediated cytotoxic autophagy by increasing dihydroceramide levels in cancer cells. Autophagy. 2021 Jun;17(6):1349-1366. doi: 10.1080/15548627.2020.1761651. Epub 2020 May 25. PMID 32397857
- [Background] Felip I, Moiola CP, Megino-Luque C, Lopez-Gil C, Cabrera S, Sole-Sanchez S, Munoz-Guardiola P, Megias-Roda E, Perez-Montoyo H, Alfon J, Yeste-Velasco M, Santacana M, Dolcet X, Reques A, Oaknin A, Rodriguez-Freixinos V, Lizcano JM, Domenech C, Gil-Moreno A, Matias-Guiu X, Colas E, Eritja N. Therapeutic potential of the new TRIB3-mediated cell autophagy anticancer drug ABTL0812 in endometrial cancer. Gynecol Oncol. 2019 May;153(2):425-435. doi: 10.1016/j.ygyno.2019.03.002. Epub 2019 Mar 7. PMID 30853360
- [Background] Lopez-Plana A, Fernandez-Nogueira P, Munoz-Guardiola P, Sole-Sanchez S, Megias-Roda E, Perez-Montoyo H, Jauregui P, Yeste-Velasco M, Gomez-Ferreria M, Erazo T, Ametller E, Recalde-Percaz L, Moragas-Garcia N, Noguera-Castells A, Mancino M, Moran T, Nadal E, Alfon J, Domenech C, Gascon P, Lizcano JM, Fuster G, Bragado P. The novel proautophagy anticancer drug ABTL0812 potentiates chemotherapy in adenocarcinoma and squamous nonsmall cell lung cancer. Int J Cancer. 2020 Aug 15;147(4):1163-1179. doi: 10.1002/ijc.32865. Epub 2020 Feb 6. PMID 31943158
- [Background] Vidal L, Victoria I, Gaba L, Martin MG, Brunet M, Colom H, Cortal M, Gomez-Ferreria M, Yeste-Velasco M, Perez A, Rodon J, Sohal DPS, Lizcano JM, Domenech C, Alfon J, Gascon P. A first-in-human phase I/Ib dose-escalation clinical trial of the autophagy inducer ABTL0812 in patients with advanced solid tumours. Eur J Cancer. 2021 Mar;146:87-94. doi: 10.1016/j.ejca.2020.12.019. Epub 2021 Feb 12. PMID 33588149
- [Background] Paris-Coderch L, Soriano A, Jimenez C, Erazo T, Munoz-Guardiola P, Masanas M, Antonelli R, Boloix A, Alfon J, Perez-Montoyo H, Yeste-Velasco M, Domenech C, Roma J, Sanchez de Toledo J, Moreno L, Lizcano JM, Gallego S, Segura MF. The antitumour drug ABTL0812 impairs neuroblastoma growth through endoplasmic reticulum stress-mediated autophagy and apoptosis. Cell Death Dis. 2020 Sep 17;11(9):773. doi: 10.1038/s41419-020-02986-w. PMID 32943619
- [Background] Mancini A, Colapietro A, Cristiano L, Rossetti A, Mattei V, Gravina GL, Perez-Montoyo H, Yeste-Velasco M, Alfon J, Domenech C, Festuccia C. Anticancer effects of ABTL0812, a clinical stage drug inducer of autophagy-mediated cancer cell death, in glioblastoma models. Front Oncol. 2022 Nov 2;12:943064. doi: 10.3389/fonc.2022.943064. eCollection 2022. PMID 36408162